CLINICAL TRIAL: NCT05175677
Title: Study of the Impact of the COVID-19 Pandemic on the Management of Type 2 Diabetic Patients in a Sample in the Paris Region
Acronym: DIABETOVID
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DIABETOVID
Record Dates: First submitted 2021-12-31; First posted 2022-01-04 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Diabetes Mellitus, Type 2
MeSH Terms: conditions — COVID-19; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Covid-19 crisis is undoubtedly the most significant event of the early 21st century. The pandemic has profoundly changed our way of life, whether as human beings, but also as patients or caregivers. This pandemic of an incredible magnitude, after having been minimized, blew a wind of fear on the whole world because of the unknown that the SARS-CoV2 virus represented. The world scientific community being destabilized, a great majority of states decided to apply a containment. In France, a strict containment was applied between March 17, 2020 and May 11, 2020 (1 month and 23 days, about 8 weeks). Diabetic and obese patients were designated as "at risk" for infection by COVID 19. Type 2 diabetes is one of the most common chronic diseases in general practice. Its regular management, we know, is largely related to lifestyle, which is particularly important in controlling the disease and preventing complications. During the first months of the pandemic, we witnessed many emergency room visits of patients with chronic pathologies, in full decompensation, due to a lack of follow-up but also due to a lack of treatment. After the first containment, in the endocrinology department of the Paris Saint-Joseph hospital, we observed that many patients had a clear imbalance of their diabetes compared to their previous history.

The main objective of this study is to show that the COVID-19 pandemic, and more precisely the strict confinement applied in France from March 17, 2020 to May 11, 2020, had an impact on diabetes control in the study population. The secondary objectives are to study the explanatory covariates via the modification of the lifestyle of diabetic patients (decrease in physical activity, increase in poor dietary habits, psychological impact related to the situation, difficulties in accessing care, modification of work arrangements).

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patients with type 2 diabetes
* Patient consulting their attending physician for the follow-up of their diabetes OR Patient consulting the GHPSJ diabetes service for the follow-up of their diabetes
* Patients who have an attending physician who follows their diabetes
* Patients living in the Paris region
* Francophone patients
* Patients who do not object to the use of their data for this research

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes, consulting between 01/09/2021 and 31/12/2021 their attending physician for the follow-up of their diabetes or the GHPSJ diabetes service for the follow-up of their diabetes who have an attending physician who follows their diabetes and living in the Paris region.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Impact on diabetes control in the study population | Month 3
  This outcome corresponds to the HbA1c levels before (3 months before March 2020) and after containment (3 months after May 2020 decontainment).

SECONDARY OUTCOMES:
Lifestyle modification for diabetic patients | Month 3
  This outcome corresponds to the weight variation before and after decontamination.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Dupuy, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Ghosal S, Sinha B, Majumder M, Misra A. Estimation of effects of nationwide lockdown for containing coronavirus infection on worsening of glycosylated haemoglobin and increase in diabetes-related complications: A simulation model using multivariate regression analysis. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):319-323. doi: 10.1016/j.dsx.2020.03.014. Epub 2020 Apr 10. PMID 32298984
- [Background] Fernandez E, Cortazar A, Bellido V. Impact of COVID-19 lockdown on glycemic control in patients with type 1 diabetes. Diabetes Res Clin Pract. 2020 Aug;166:108348. doi: 10.1016/j.diabres.2020.108348. Epub 2020 Jul 22. PMID 32711000
- [Background] Ruiz-Roso MB, Knott-Torcal C, Matilla-Escalante DC, Garcimartin A, Sampedro-Nunez MA, Davalos A, Marazuela M. COVID-19 Lockdown and Changes of the Dietary Pattern and Physical Activity Habits in a Cohort of Patients with Type 2 Diabetes Mellitus. Nutrients. 2020 Aug 4;12(8):2327. doi: 10.3390/nu12082327. PMID 32759636
- [Background] Ruissen MM, Regeer H, Landstra CP, Schroijen M, Jazet I, Nijhoff MF, Pijl H, Ballieux BEPB, Dekkers O, Huisman SD, de Koning EJP. Increased stress, weight gain and less exercise in relation to glycemic control in people with type 1 and type 2 diabetes during the COVID-19 pandemic. BMJ Open Diabetes Res Care. 2021 Jan;9(1):e002035. doi: 10.1136/bmjdrc-2020-002035. PMID 33431602
- [Background] Karatas S, Yesim T, Beysel S. Impact of lockdown COVID-19 on metabolic control in type 2 diabetes mellitus and healthy people. Prim Care Diabetes. 2021 Jun;15(3):424-427. doi: 10.1016/j.pcd.2021.01.003. Epub 2021 Jan 9. PMID 33441263
- [Background] Tanji Y, Sawada S, Watanabe T, Mita T, Kobayashi Y, Murakami T, Metoki H, Akai H. Impact of COVID-19 pandemic on glycemic control among outpatients with type 2 diabetes in Japan: A hospital-based survey from a country without lockdown. Diabetes Res Clin Pract. 2021 Jun;176:108840. doi: 10.1016/j.diabres.2021.108840. Epub 2021 Apr 30. PMID 33933499